CLINICAL TRIAL: NCT02642666
Title: The Effects of Yoga on Attention, Impulsivity and Hyperactivity in Pre-school Age Children With ADHD Symptoms
Brief Title: The Effects of Yoga on Attention, Impulsivity and Hyperactivity in Pre-school Age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 801230
Record Dates: First submitted 2015-12-23; First posted 2015-12-30 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: ADHD
Keywords: Attention; Hyperactivity; Impulsivity; Yoga; Preschool
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm; Impulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga intervention (Experimental): While in the yoga intervention arm of the study participants will practice yoga at home and at school for six weeks with the goal of practicing yoga daily during that time period. Yoga classes will be held twice a week at school. On the days that the children do not practice yoga at school, they will practice yoga at home with the use of a children's yoga video that mirrors the yoga class that they attend at school.
  Interventions: Behavioral: Children's Yoga
- Normal school and home activities (No Intervention): While in the wait-list group the children will continue with their regular activities both at home and at school.

INTERVENTIONS:
Behavioral: Children's Yoga — Trained children's yoga instructors will guide the children through 30 minute yoga classes (in-person and on the yoga video), using a manualized curriculum from If I Was a Bird Yoga ™ with child centered themes. Each class will have a similar structure, set of poses, and breathing exercises, but the theme of the class will change every two weeks. The themes for the classes are "ocean yoga adventure", "jungle yoga adventure" and "outer space yoga adventure". The study participants will spend two weeks practicing the same theme at home and at school before moving on to the next theme.
  Arms: Yoga intervention

SUMMARY:
This pilot project will evaluate yoga as an intervention to improve attention and reduce challenging behaviors such as hyperactivity and impulsivity, rated by parent and teachers, in preschool age children with or "at risk" for attention-deficit hyperactivity disorder (ADHD). "At Risk" for ADHD will be defined as four or more hyperactive/impulsive and/or inattentive symptoms on the ADHD Rating Scale IV-Preschool Version as rated by parents or teachers. Using a randomized wait-list controlled experimental design, the investigators will explore the efficacy of practicing yoga for 6 weeks on behavioral symptoms, attentional control using a computer based tasks of attention, and heart rate variability (HRV), which is a measure of self-regulatory capacity. The investigators hypothesize that practicing yoga for six weeks of will improve ADHD and other behavioral symptoms based on parent and teacher rating scales, which will correlate with improvements in scores on the computer based task of attention as well as with improvements in HRV.

DETAILED DESCRIPTION:
Background: Symptoms of attention-deficit hyperactivity disorder (ADHD) are often observable by preschool age and can be associated with similar behavioral, social, and cognitive impairments as seen in older children with ADHD. Seventy to eighty percent of preschoolers with symptoms of ADHD continue to display these symptoms in elementary school. Behavioral therapies are recommended as first line treatments in this age group. There have been some small but promising studies looking at yoga as an intervention for school age children with ADHD, but none have looked specifically at yoga as an intervention for preschool age children with ADHD symptoms (Birdee et al, 2009).

Objective: To determine if yoga improves hyperactive/impulsive symptoms and attention in preschool age children with or "at risk" for ADHD.

Study design: A randomized wait-list controlled trial exploring whether 6 weeks of children's yoga improves behavioral symptoms, task-related scores of attention, and increases heart rate variability in preschool age children "at risk" for or diagnosed with ADHD. The investigators plan to enroll a total of 30 children ages 3-5 years old. "At risk" for ADHD will be defined as four or more inattentive or hyperactive/impulsive symptoms rated by parents and teachers on the ADHD Rating Scale-IV Preschool Version.

Procedures: The investigators will evaluate the efficacy of yoga for improving ADHD and other behavioral symptoms using parent and teacher rating scales (ADHD Rating Scale-IV Preschool Version; Strengths and Difficulties Questionnaire), as well as objective measures including computer based tasks of attention and executive function (KiTAP, Test of Attentional Performance for Children), and heart rate variability (HRV), a physiologic measure of self-regulatory capacity. HRV will be assessed during an active, attention computer task (using the emWave ® desktop device), as well as during a relaxed state, in a breathing exercise paired with verbal affirmations. The protocol includes baseline, post-treatment and 3 month follow-up assessments. The intervention consists of school and home yoga sessions. School sessions will be held twice a week at Triumph Center for Early Childhood Education, which is a local preschool associated with University of California, Davis. The school based yoga classes will be lead by trained child yoga instructors using a manualized yoga protocol that is 30 minute long. Home session will include use of a children's yoga video featuring the same protocol to practice at home on the days that the children do not participate at school. The goal is for daily yoga practice during the 6 week intervention period. Home yoga practice will be documented daily by parents completing a brief online survey that is emailed to them. Generalization of the skills learned during the yoga sessions to behaviorally-challenging situations will be specifically developed by teaching the parents and teachers to "cue" the children to integrate skills learned in the yoga sessions into their daily routine. The goal is for the children to learn to use breathing practices and affirmations to help regain calmness and focus when their behaviors become challenging. A questionnaire will assess parent and teacher perception regarding the use of yoga in the children's daily life, its effect on challenging behaviors, and their satisfaction with the intervention. Optional focus groups will also be done with the parents and teachers of the children who participate in the study in order to gather qualitative data about the yoga intervention.

Statistical Methods and Power Analysis: Outcome distributions will be visualized and, if necessary, log-transformed to reduce skewness or stabilize variances. For this wait-list design, the primary assessment of treatment effects will be estimated by comparing treatment and control groups on baseline-adjusted mean outcomes at the first follow-up and reported with 95% Confidence Intervals. Between- and within-group contrasts involving outcomes at the 2nd follow-up time will permit exploration of treatment durability. The primary index of HRV will be the standard deviation of beat-to-beat intervals, but other time- and frequency-domain indices will be evaluated in exploratory analyses. Assuming pre/post correlations of 60%, our target sample size of 30 subjects will permit estimating treatment effects with margins of error of 0.41 standard deviations and provide 80% power (with 2-sided alpha=5%) to detect between-group effects as small as 0.59 standard deviations.

Gaps in knowledge: The majority of the studies on yoga for children with ADHD have been conducted in school aged children, and only one was completed in the United States. None have looked specifically at yoga as an intervention for ADHD symptoms in preschoolers. In addition, none of these studies included physiologic measures such as vagal tone, which has been shown to increase in adults who practice yoga. Physiologic measures are valuable because they are an objective measure of treatment response, may give evidence to support the role, and perhaps mechanism by which yoga may affect change in ADHD. The investigators will assess heart rate variability (HRV), a measure of the beat-to-beat changes in heart rate, which reflects the activity of the vagus nerve, a key component of the parasympathetic nervous system, which mediates changes in heart rate. Reduced HRV is associated with increased morbidity and mortality, while increased HRV is associated with physiologic resiliency, the ability to self-regulate and improved performance on tasks of executive function. Compared to healthy controls, children with ADHD have higher mean heart rates, and unmedicated children have significantly decreased HRV. In adults, HRV has been found to increase in response to both exercise and biofeedback. A study in children with ADHD evaluated the use of biofeedback using HRV coherence, synchronization of the heart rhythm pattern, and found that it improved cognitive function and behaviors. HRV has not been evaluated in relation to yoga training in young children with ADHD symptoms.

Innovation: This project is novel in its subject population, preschoolers, teaching of yoga at the school, use of manualized treatments, objective measures and wait-list randomized control methodology. While there are many studies in exercise, yoga and meditation for children, many lack sophisticated methodology to guide clinical practice. The proposed methods are not highly innovative, but they are critical to moving the field forward and providing direction to clinicians, parents and teachers in need of research to guide their clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* English speaking children
* Ages of 3-5 years old
* Diagnosed with ADHD or "at risk" for ADHD (defined as four or more hyperactive/impulsive and/or inattentive symptoms on the ADHD Rating Scale IV-Preschool Version rated by parents or teachers)

  * The yoga intervention will be given in addition to any other behavioral and/or medication treatments that the study participants are receiving. We will document any medications or behavioral therapies that participants are on during the study.
* The child's parent agrees to support their child in doing home yoga practice using a yoga video, which may range from being present and giving verbal encouragement to their child but not engaging in the yoga themselves (which is recommended and preferred for pregnant women) to practicing yoga along with their child using the yoga videos based on the parent's preference and comfort level with practicing yoga.
* Children with common co-morbid diagnoses such as autism spectrum disorder, anxiety, oppositional defiant disorder, and learning differences.
* Children's parents and teachers (including pregnant women if applicable) will be included in the study, as they will be asked to complete study questionnaires and surveys.

Exclusion Criteria:

* Non-English speaking children
* Children who have a medical condition or physical impairment precluding them from safely exercising and participating in the yoga classes (eg. spastic quadriplegic cerebral palsy, critical congenital heart disease, uncontrolled asthma, uncontrolled seizure disorder, etc.).
* Adults unable to consent
* Children younger than 3 or older than 5 at the start of the study intervention
* Prisoners

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in ADHD Rating Scale-IV Preschool Version Scores | Baseline, after the first six week yoga intervention, after the second six week yoga intervention, 3 month follow up
  An 18 item questionnaire with reliable, valid and developmentally appropriate statements based on ADHD symptoms defined by the Diagnostic and Statistical Manual (DSM)-IV-Text Revision. Parents and teachers will be asked to rate the frequency of the behaviors listed. It will be used for screening and monitoring response to the intervention.
Change in Strengths and Difficulties Questionnaire Scores | Baseline, after the first six week yoga intervention, after the second six week yoga intervention, 3 month follow up
  A 30 item questionnaire validated with five sub-scales: Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention Symptoms, Peer Problems and Pro-social Behaviors. There is a total difficulty score, and a pro-social scale score. Both parents and teachers will be asked to complete this questionnaire. It will be used for screening and monitoring response to the intervention.
Change in KiTAP Test of Attentional Performance for Children Scores | Baseline, after the first six week yoga intervention, after the second six week yoga intervention, 3 month follow up
  The KiTAP is a computer administered child-friendly test with the theme of an enchanted castle. Four of the 8 sub-tests (alertness, distractibility, flexibility, and go/no-go) are feasible and reliable for a mental age of 3 years and higher, and correlated with behavioral ratings of hyperactivity and attention. The investigators will collect percent correct and response time on the 4 sub-tests to assess attention and executive function.
Change in Heart rate variability (HRV) | Baseline, after the first six week yoga intervention, after the second six week yoga intervention, 3 month follow up
  HRV will be measures using the emWave® Coherence System by HeartMath. The emWave®, which is a commercially available device, is a photoplethysmography optical sensor (similar to a pulse ox) that will be placed on the subjects earlobe to measure the beat-to-beat changes in heart rate, which constitutes HRV. A computer program interprets the inter-beat-intervals into a spectral display of the heart rhythm patterns. HRV will be measured during the KiTAP test of attention/executive function and during a yogic breathing exercise paired with verbal affirmations.

SECONDARY OUTCOMES:
Change in Likert scale of "Time on Task" during group yoga classes | During the six week intervention, after the school based yoga classes
  A seven point Likert scale rated by the yoga instructor will be completed for each study participant after each school based yoga class.
Change in Strategies Used to Address Challenging Behaviors | Baseline, after the first six week yoga intervention, after the second six week yoga intervention, 3 month follow up
  A three item questionnaire for parents and teachers about the strategies they use to address challenging behaviors in their child or student. For each strategy they use they are asked to rate how well it works on a semantic differential scale from "Ineffective" to "Very effective", and if their child/student is receptive to using the strategy.
Parent and Teacher Satisfaction Questionnaire | After 6 to 12 weeks
  A 7 to 9 item questionnaire to assess the feasibility of the intervention by assessing parent and teacher satisfaction with the intervention and their perception about how challenging it was to implement.
Parent and Teacher Perception Questionnaire | After 6 to 12 weeks
  A 12-14 item questionnaire to assess parent and teacher perceptions about such things as the usefulness of the yoga breathing exercises, details about the children's behavior not addressed in the rating scales, ease of use of the yoga video for parents, and duration of effects after practicing yoga.
Feasibility | Through study completion, an average of 18 weeks
  The investigators will assess the feasibility of the intervention by assessing drop-out rates.
Qualitative Data About the Feasibility of the Yoga Intervention Using Focus Group Discussions with Parents and Teachers | After 6 to 12 weeks
  Parents and teachers will be invited to participate in a focus group discussion about their perception of their child's/student's experience during the yoga intervention. The parent and teacher focus groups will be held separately and consist of 4 to 6 questions that will take about 20-30 minutes to discuss. The discussions will be record, and then transcribed and coded. The focus group questions will help to gain detailed qualitative data about parent and teacher perceptions about such things as the usefulness of the yoga breathing exercises, descriptions of the changes in children's behavior that were noticed during the yoga intervention (included any changes in sleep, appetite and overall behavior), how long the effects of practicing yoga seemed to last, ease of use of the yoga video for parents, and effects on parent and teacher stress levels during the yoga intervention.
Measure of Adherence with Home Yoga Practice | Through study completion, an average of 18 weeks
  The investigators will assess the number of home based sessions each child participated in to assess adherence with the program. Home based yoga sessions will be tracked in REDCap using parent's responses to the daily emails they receive. For parents who don't have easy access to email a hard copy of the Daily Survey to Assess Frequency of Yoga Practice will be sent home for parents to complete each week.
Measure of Adherence with School Yoga Practice | Through study completion, an average of 18 weeks
  The investigators will assess the number of school based sessions each child participated in to assess adherence with the program. Attendance at school based yoga session will be tracked by the yoga instructors.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha C Cohen, MD, Principal Investigator — University of California, Davis
Locations (1):
- Triumph Center for Early Childhood Education, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participants data will be de-identified and analyzed as a group.

REFERENCES:
- [Background] Barkley RA. Attention-Deficit Hyperactivity Disorder. Fourth Edition ed. Barkley RA, editor. New York, NY: The Guilford Press; 2015.
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Molina BSG, Hinshaw SP, Swanson JM, Arnold LE, Vitiello B, Jensen PS, Epstein JN, Hoza B, Hechtman L, Abikoff HB, Elliott GR, Greenhill LL, Newcorn JH, Wells KC, Wigal T, Gibbons RD, Hur K, Houck PR; MTA Cooperative Group. The MTA at 8 years: prospective follow-up of children treated for combined-type ADHD in a multisite study. J Am Acad Child Adolesc Psychiatry. 2009 May;48(5):484-500. doi: 10.1097/CHI.0b013e31819c23d0. PMID 19318991
- [Background] Knox A, Schneider A, Abucayan F, Hervey C, Tran C, Hessl D, Berry-Kravis E. Feasibility, reliability, and clinical validity of the Test of Attentional Performance for Children (KiTAP) in Fragile X syndrome (FXS). J Neurodev Disord. 2012 Feb 8;4(1):2. doi: 10.1186/1866-1955-4-2. PMID 22958782
- [Background] McCraty R, Shaffer F. Heart Rate Variability: New Perspectives on Physiological Mechanisms, Assessment of Self-regulatory Capacity, and Health risk. Glob Adv Health Med. 2015 Jan;4(1):46-61. doi: 10.7453/gahmj.2014.073. PMID 25694852
- [Background] Buchhorn R, Conzelmann A, Willaschek C, Stork D, Taurines R, Renner TJ. Heart rate variability and methylphenidate in children with ADHD. Atten Defic Hyperact Disord. 2012 Jun;4(2):85-91. doi: 10.1007/s12402-012-0072-8. Epub 2012 Feb 11. PMID 22328340
- [Background] Jensen PS, Kenny DT. The effects of yoga on the attention and behavior of boys with Attention-Deficit/ hyperactivity Disorder (ADHD). J Atten Disord. 2004 May;7(4):205-16. doi: 10.1177/108705470400700403. PMID 15487477
- [Background] Haffner J, Roos J, Goldstein N, Parzer P, Resch F. [The effectiveness of body-oriented methods of therapy in the treatment of attention-deficit hyperactivity disorder (ADHD): results of a controlled pilot study]. Z Kinder Jugendpsychiatr Psychother. 2006 Jan;34(1):37-47. doi: 10.1024/1422-4917.34.1.37. German. PMID 16485612
- [Background] Peck HL, Kehle TJ, Bray MA, Theodore LA. Yoga as an Intervention for Children With Attention Problems. School Psychology Review. 2005;34(3):415.
- [Background] Harrison LJ. Sahaja Yoga Meditation as a Family Treatment Program for Children with Attention Deficit-Hyperactivity Disorder. Clinical Child Psychology and Psychiatry. 2004; 9(4):479-97.
- [Background] Hariprasad VR, Arasappa R, Varambally S, Srinath S, Gangadhar BN. Feasibility and efficacy of yoga as an add-on intervention in attention deficit-hyperactivity disorder: An exploratory study. Indian J Psychiatry. 2013 Jul;55(Suppl 3):S379-84. doi: 10.4103/0019-5545.116317. PMID 24049203
- [Background] Balasubramaniam M, Telles S, Doraiswamy PM. Yoga on our minds: a systematic review of yoga for neuropsychiatric disorders. Front Psychiatry. 2013 Jan 25;3:117. doi: 10.3389/fpsyt.2012.00117. eCollection 2012. PMID 23355825
- [Background] Schmalzl L, Powers C, Henje Blom E. Neurophysiological and neurocognitive mechanisms underlying the effects of yoga-based practices: towards a comprehensive theoretical framework. Front Hum Neurosci. 2015 May 8;9:235. doi: 10.3389/fnhum.2015.00235. eCollection 2015. PMID 26005409
- [Background] Birdee GS, Yeh GY, Wayne PM, Phillips RS, Davis RB, Gardiner P. Clinical applications of yoga for the pediatric population: a systematic review. Acad Pediatr. 2009 Jul-Aug;9(4):212-220.e1-9. doi: 10.1016/j.acap.2009.04.002. PMID 19608122
- [Background] Prinsloo GE, Rauch HG, Derman WE. A brief review and clinical application of heart rate variability biofeedback in sports, exercise, and rehabilitation medicine. Phys Sportsmed. 2014 May;42(2):88-99. doi: 10.3810/psm.2014.05.2061. PMID 24875976
- [Background] Lloyd A, Brett D, Wesnes K. Coherence training in children with attention-deficit hyperactivity disorder: cognitive functions and behavioral changes. Altern Ther Health Med. 2010 Jul-Aug;16(4):34-42. PMID 20653294
- [Background] Van Breukelen GJ. ANCOVA versus change from baseline: more power in randomized studies, more bias in nonrandomized studies [corrected]. J Clin Epidemiol. 2006 Sep;59(9):920-5. doi: 10.1016/j.jclinepi.2006.02.007. Epub 2006 Jun 23. PMID 16895814
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Berwid OG, Halperin JM. Emerging support for a role of exercise in attention-deficit/hyperactivity disorder intervention planning. Curr Psychiatry Rep. 2012 Oct;14(5):543-51. doi: 10.1007/s11920-012-0297-4. PMID 22895892
- [Background] Subcommittee on Attention-Deficit/Hyperactivity Disorder; Steering Committee on Quality Improvement and Management; Wolraich M, Brown L, Brown RT, DuPaul G, Earls M, Feldman HM, Ganiats TG, Kaplanek B, Meyer B, Perrin J, Pierce K, Reiff M, Stein MT, Visser S. ADHD: clinical practice guideline for the diagnosis, evaluation, and treatment of attention-deficit/hyperactivity disorder in children and adolescents. Pediatrics. 2011 Nov;128(5):1007-22. doi: 10.1542/peds.2011-2654. Epub 2011 Oct 16. PMID 22003063
- [Background] Halperin JM, Marks DJ, Bedard AC, Chacko A, Curchack JT, Yoon CA, Healey DM. Training executive, attention, and motor skills: a proof-of-concept study in preschool children With ADHD. J Atten Disord. 2013 Nov;17(8):711-21. doi: 10.1177/1087054711435681. Epub 2012 Mar 5. PMID 22392551
- [Background] Krisanaprakornkit T, Ngamjarus C, Witoonchart C, Piyavhatkul N. Meditation therapies for attention-deficit/hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD006507. doi: 10.1002/14651858.CD006507.pub2. PMID 20556767